CLINICAL TRIAL: NCT00693004
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of PRX-03140 as Monotherapy in Subjects With Alzheimer's Disease
Brief Title: Study of PRX-03140 Monotherapy in Subjects With Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Epix Pharmaceuticals, Inc. (Industry)
Responsible Party: Elkan R. Gamzu, PhD, EPIX Pharmaceuticals, Inc.
Purpose: Treatment
Other Study IDs: Protocol 03140-203
Record Dates: First submitted 2008-05-30; First posted 2008-06-06 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PRX-03140 (Experimental)
  Interventions: Drug: PRX-03140
- donepezil (Active Comparator)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: PRX-03140
  Arms: PRX-03140
Drug: Donepezil
  Arms: donepezil
Drug: Placebo
  Arms: Placebo

SUMMARY:
A randomized placebo-controlled study to evaluate the efficacy of PRX-03140 monotherapy in subjects with Alzheimer's disease. The study consists of a 3-month double-blind treatment period and an optional 3-month extension period.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women with a clinical diagnosis of Probable AD
* MMSE score 16 to 24 inclusive
* Age >50 and <90 years
* Brain CT or MRI scan Consistent with a primary diagnosis of AD within 12 months
* Neurological examination without focal deficits (excluding changes attributable to peripheral nervous system disease, trauma or congenital birth deficits)
* No history or evidence of any other CNS disorder that could be interpreted as a cause of dementia
* No diagnosis of vascular dementia
* No history of significant psychiatric illness such as schizophrenia or bipolar affective disorder. Subjects with major depressive disorder on a stable dose of an antidepressant for >6 months may be eligible
* No evidence of the following: current vitamin B12 deficiency, positive syphilis serology, positive HIV test, or abnormalities in thyroid function
* No cognitive rehabilitation within 6 months of the study
* Subject has a regular caregiver willing to attend all study visits
* Signed informed consent by the subject (and legal guardian, if applicable)

Exclusion Criteria:

* No history of drug or alcohol abuse
* No clinically significant laboratory abnormalities or medical history
* No investigational drug within 30 days of Randomization
* Intolerance or allergy to cholinesterase inhibitors
* Cannot have been on cholinesterase inhibitors for AD for > 2 years
* If have been on cholinesterase inhibitors for < 2 years, must have been discontinued >= 2 months prior to randomization
* Cannot have received memantine within 2 months
* No clinically significant ECG abnormalities prior to randomization
* No history of uncontrolled seizure disorder within 12 months
* Cannot be taking MAO inhibitors, bupropion,fluoxetine, paroxetine, quinidine
* No history of malignancy within 3 years of randomization
* Women cannot be pregnant or breastfeeding

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive subscale.

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Barrow Neurological Institute, Phoenix, Arizona
  - PsyPharma Clinical Research, Inc., Phoenix, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - Synergy Clinical Research Center, National City, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Torrance Clinical Research, Torrance, California
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Compass Research, Orlando, Florida
  - Berma Research Group, Plantation, Florida
  - Meridien Research, St. Petersburg, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Roskamp Institute, Tampa, Florida
  - Four Rivers Clinical Research, Paducah, Kentucky
  - J. Gary Booker, MD, APMC, Shreveport, Louisiana
  - Maine Neurology, Scarborough, Maine
  - The ICPS Group, Norwood, Massachusetts
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - Global Medical Institutes, Princeton, New Jersey
  - Social Psychiatry Research Institute, Brooklyn, New York
  - The Mount Sinai Medical Center, New York, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - The Neurological Institute, P.A., Charlotte, North Carolina
  - MedArk, Morgantown, North Carolina
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Todd Swick, MD, PA, Houston, Texas
  - The Memory Clinic, Bennington, Vermont
  - The Glennan Center for Geriatrics & Gerontology, Eastern Virginia Medical School, Norfolk, Virginia
  - The Center for Excellence in Aging and Geriatric Health, Williamsburg, Virginia